

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

A Pilot Study of StrataXRT, a Topical Silicone Barrier, to Prevent Auricular Radiation Dermatitis in Pediatric Patients Undergoing Proton Cerebrospinal Radiation Therapy 2018-0980

| Study Chair: Susan L. McGovern | |
|--------------------------------|-----------------------|
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

#### STUDY SUMMARY

If you are reading and signing this form on behalf of a potential participant, please note: Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

The goal of this research study is to learn if a type of ointment called StrataXRT can safely and effectively help to prevent radiation dermatitis (skin burns and side effects caused by radiation) in children receiving craniospinal irradiation (CSI), a type of proton therapy radiation.

In this study, StrataXRT will be compared to a placebo. A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with StrataXRT to learn if StrataXRT has any real effect.

StrataXRT is FDA approved and commercially available for treatment of radiation dermatitis in adult populations receiving photon radiation therapy. Its use in this study is investigational.

StrataXRT may help prevent or decrease severe skin rash, pain, itching, skin peeling, and dry skin from CSI. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment.

You can read a full list of potential side effects below in the Possible Risks section of this consent.

You may use StrataXRT/placebo during radiation for up to 6 weeks...

StrataXRT/placebo will be provided at no cost to you. You and/or your insurance provider will be responsible for the cost of radiation therapy.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive standard photon radiation therapy outside of this study. You may choose to receive other investigational therapy, if available. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

### 1. STUDY DETAILS

Up to 30 participants will be enrolled in this study. All will take part at MD Anderson.

If you agree to take part in this study, you will be given a placebo and StrataXRT. The placebo will be placed on one ear and StrataXRT will be applied to the other. However neither you nor the study doctor will know which ear has been treated with placebo and which has been treated with StrataXRT.

The research team will show you how to apply the ointments from the forehead to behind the ears. You will begin applying the ointments 2 times every day, about 12 hours apart (1 time in the morning, 1 time in the evening) on the first day of radiation therapy and continue every day until the last day of radiation therapy (about 6 weeks). It is very important you apply the same ointment to the same ear each time, about 15 minutes before each radiation treatment.

You will be given an application journal to write down when you apply the morning and evening applications of the ointments.

If you have side effects, you may be given standard medications (such as Aquaphor, Coolmagic, Meiplex, or Silvadene) to help reduce or prevent side effects. Talk with the study staff about these medications and how they are given, including their risks.

#### **Study Visits**

At the time that you sign this consent (baseline) and every week for up to 7 weeks, you will complete a questionnaire about your skin-related symptoms. Additionally, pictures of your forehead and ears will be taken.

You will no longer be able to use StrataXRT/placebo if the side effects get worse, if intolerable side effects occur, or if you are unable to follow study directions. Your

participation in this study will be over after you have completed radiation therapy and your final treatment completion visit.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The known side effects are listed in this form, but they will vary from person to person.

At this time, there are no known risks for **StrataXRT**.

You will receive a standard consent document that will describe the risks of **proton** beam therapy (the standard-of-care treatment).

### Other Risks

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaire, you are encouraged to contact your doctor or the study chair.

This study may involve unpredictable risks to the participants.

### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-2933 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

- 4. You may ask the study chair (Dr. Susan L. McGovern, at 713-563-2300) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-2933 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.

# **Future Research**

Your personal information is being collected as part of this study. This information, or data, may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

Before being shared for future research, every effort will be made to remove your identifying information from any data. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

# **Authorization for Use and Disclosure of Protected Health Information (PHI):**

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

If photographs taken during this study are published, steps will be taken to protect your identity.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

| I understand the information in this consent form. I have had a character consent form for this study, or have had it read to me. I have had a about it, ask questions, and talk about it with others as needed. I gi permission to enroll me on this study. By signing this consent form any of my legal rights. I will be given a signed copy of this consent | chance to think<br>ive the study chair<br>, I am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| LEGALLY AUTHORIZED REPRESENTATIVE (LAR) The following signature line should only be filled out when the parti the capacity to legally consent to take part in the study and/or sign or her own behalf. | |
| SIGNATURE OF LAR | DATE |
| RELATIONSHIP TO PARTICIPANT WITNESS TO CONSENT I was present during the explanation of the research to be performe 2018-0980. | ed under Protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT<br>PRESENTATION (OTHER THAN PHYSICIAN OR STUDY<br>CHAIR) | DATE |
| A witness signature is only required for vulnerable adult participant witnessing the assent of a pediatric participant, leave this line blank the witness to assent page instead. | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his representative, using language that is understandable and appropr have fully informed this participant of the nature of this study and its and risks and that the participant understood this explanation. | iate. I believe that I |
| PERSON OBTAINING CONSENT | DATE |

# PARENT/GUARDIAN PERMISSION I have read and understand the description of this research. I have had a chance to discuss the study and ask questions. My questions have been answered. I give permission for my child or ward to take part in this study. SIGNATURE OF PARENT/GUARDIAN DATE DATE SIGNATURE OF PARENT/GUARDIAN Signature of Other Parent (Optional, unless required by the IRB.) The IRB has determined that the signature of both parents is required. If not obtaining both parental signatures, please indicate reason below: Other parent is deceased, unknown, incompetent, or not reasonably available. Parent/Guardian signing above has sole legal responsibility for the care and custody of the child. **X** The IRB has determined that the signature of both parents is NOT required. WITNESS TO PARENTAL/GUARDIAN PERMISSION I was present during the explanation of the research to be performed under Protocol 2018-0980. The child participant was also present. In my opinion, the parent(s)/guardian provided permission for the child to participate in the research.

SIGNATURE OF WITNESS TO THE PARENTAL/GUARDIAN

PERMISSION (OTHER THAN PARENT/GUARDIAN OR

MEMBER OF THE STUDY TEAM)

DATE

# **ASSENT OF MINOR**

(Entire section must be completed if the participant's intellectual age is at least 7 and less than 18 years. Participants with an intellectual age of 7 - 12 are not required to sign.)

| If written assent is not obtained on an age-appropriate participant, check renot: | eason why |
|---|---|
| 1.) The participant's intellectual age is less than seven. | |
| 2.) The participant dissented, but the participant's parent(s)/guardia intervention(s) or procedure(s) involved in the research hold out possibility of a direct benefit that is important to the health and/o of the participant and is available only in the context of this rese | the<br>or well being |
| 3.) Other: | |
| I have been told what I will be asked to do in this study. | |
| I have been told that I do not have to be in this study. If I decide not to be in this study, no one will be mad at me. I may quit at any time, but if I do, I may need to take a different treatment. | |
| I have had a chance to talk about the study and ask the study doctor ques my questions have been answered. I agree to be in this study and do what to do so long as I want to stay in this study. I agree that the study doctor of this study. By signing this paper, I am not giving up any of my legal rights. given a copy of this document. | at I am asked<br>can put me on |
| SIGNATURE OF MINOR (Age 13-17) | DATE |
| WITNESS TO ASSENT I was present during the explanation of the research to be performed unde 2018-0980. The child participant was also present. In my opinion, the chi to participate in the research. (Note: If obtaining assent, a witness signature required.) | ld assented |
| SIGNATURE OF WITNESS TO THE ASSENT (OTHER THAN PARENT/GUARDIAN OR MEMBER OF THE STUDY TEAM) | DATE |

# **TRANSLATOR**

| subtractions) into | med consent as written (without additions orand assisted the people of Language) | |
|---|---|---|
| `` | by translating all questions and respo | onses during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| ☐ Please check here if the translator was a member of the research team. (If checked, a witness, other than the translator, must sign the witness line below.) | | |
| SIGNATURE OF WITNESS TO (OTHER THAN TRANSLATOR, I | | DATE |